CLINICAL TRIAL: NCT03682042
Title: A Cluster Randomized Clinical Trial of Umbilical Cord Milking Versus Early Cord Clamping on Short and Long-term Outcomes in Neonates Who Are Non-Vigorous at Birth
Brief Title: Comparative Outcomes Related to Delivery-room Cord Milking In Low-resourced Kountries Developmental Follow Up
Acronym: CORDMILK-FU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Sharp HealthCare (Other); Thomas Jefferson University (Other); University of California, San Diego (Other); St. Louis University (Other); KLE Academy of Higher Education and Research (Deemed- to- be-University), Jawaharlal Nehru Medical College (JNMC), Belagavi, India (Unknown); Government Medical College, Nagpur (Industry); Daga Memorial Maternity and Children's Hospital, Nagpur, India (Unknown); Mahatma Gandhi Institute of Medical Sciences/ Kasturba Hospital, Wardha, India (Unknown); Karnataka Institute of Medical Sciences, Hubbali, India (Unknown); All India Institute of Medical Sciences (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Indira Gandhi Government Medical College & Hospital, Nagpur, India (Unknown); Pimpri Chinchwad Municipal Corporation's Post-Graduate Institute, Yashwantrao Chavan Memorial Hospital, Pune, India (Unknown)
Responsible Party: Principal Investigator, Zubair Aghai, Professor of Pediatrics, Nemours Children's Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CORDMILK FU; R01HD102967 (NIH)
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Birth Asphyxia
Keywords: Placental transfusion
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Asphyxia Neonatorum; Fetofetal Transfusion | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: Neurodevelopmental assessments will be done at 2 years of age (22-26 months) for subjects who were randomized to receive either early cord clamping or umbilical cord milking as part of the CORDMILK trial.
Who Masked: Outcomes Assessor
Masking Description: Neurodevelopmental providers will be blinded to the randomization of the toddler during the examination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical Cord Milking (Active Comparator): At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped. This procedure infuses a placental transfusion of blood into the infant and can be done in 10-15 seconds.
  Interventions: Other: Umbilical Cord Milking
- Early Cord Clamping (No Intervention): The umbilical cord is clamped immediately after the delivery (within 60 seconds).

INTERVENTIONS:
Other: Umbilical Cord Milking — At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped. This procedure infuses a placental transfusion of blood into the infant and can be done in 10-15 seconds.
  Arms: Umbilical Cord Milking

SUMMARY:
An extension of the CORDMILK trial, the CORDMILK follow-up trial will evaluate the neurodevelopmental outcomes at 22-26 months age of term/late preterm infants who were non-vigorous at birth and received umbilical cord milking (UCM) or early cord clamping (ECC).

DETAILED DESCRIPTION:
The CORDMILK Follow-up trial will examine the difference in survival and neurodevelopmental impairment of infants who were non-vigorous at birth and enrolled in the CORDMILK trial. The difference in survival and neurodevelopmental impairment in infants who received UCM and ECC will be assessed using standardized neurological and developmental assessment tools at 22-26 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in CORDMILK trial
* Non-vigorous at birth

Exclusion Criteria:

* None

Ages: 22 Months to 26 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3442 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopmental Outcome at 2 Years of Age | 22-26 months
  Neurodevelopmental assessment will be performed by the trained and experienced examiner who will be blinded to the interventions.
  Severe neurodevelopmental impairment will be defined having at least one of the following: BSID (IV) composite cognitive score <70, GMFCS level 3-5, blindness (vision <20/200), or hearing impairment requiring hearing aids/cochlear implant. Moderate neurodevelopmental impairment will be defined as having a cognitive composite score 70-84, GMFCS level 2, unilateral blindness (vision/20/200 in only one eye), or hearing impairment with no amplification/cochlear implant.

SECONDARY OUTCOMES:
Neurodevelopmental Outcome at 1 Year of Age | 10-14 months
  Neurodevelopmental assessment will be performed by the trained and experienced examiner who will be blinded to the intervention using the Developmental Assessment Scales for Indian Infants (DASII). DAASI provides developmental motor quotient (DMoQ), developmental mental quotient (DMeQ), and composite developmental quotient (DQ). With a mean DQ of 100 and standard deviation (SD) of 15, 1SD and 2SD below mean correspond to DQ of 85 and 70, respectively. A DMoQ, DMeQ or DQ score of <70 (2SD) is considered as neurodevelopmental impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Zubair Aghai, MD, Principal Investigator — Nemours Children's Clinic; Anup Katheria, MD, Principal Investigator — Sharp Mary Birch Hospital for Women & Newborns; Sangappa Dhaded, Principal Investigator — KLE Academy of Higher Education and Research
Locations (9):
- India (9):
  - KLE Academy of Higher Education and Research (Deemed-to-be-University) Jawaharlal Nehru Medical College, Belagavi, Karnataka
  - Indira Gandhi Government Medical College & Hospital, Nagpur, Maharashtra
  - Pimpri Chinchwad Municipal Corporation's Post-Graduate Institute, Yashwantrao Chavan Memorial Hospital, Pune, Maharashtra
  - Government Medical College, Chandrapur, MS
  - Daga Memorial Woman and Children Hospital, Nagpur, MS
  - Government Medical College and Hospital, Nagpur, MS
  - All India Institute of Medical Science, Nagpur, MS
  - Mahatma Gandhi Institute of Medical Sciences/ Kasturba Hospital, Wardha, MS
  - Sawai Man Singh (SMS) Medical College, Jaipur, Rajasthan

REFERENCES:
- [Derived] Yogeshkumar S, Vernekar SS, Dhaded SM, Talekar K, Leiby BE, Hartman R, Vaucher Y, Chouthai N, Girish M, Jain M, Jain S, Parvekar S, Jain V, Patankar A, Suryawanshi M, Tiwari M, Waikar M, Nashine N, Ambike D, Asalkar M, Kulkarni R, Haribhaktha S, Narkhede H, Chaudhari S, Kamble M, Shrirame D, Falke B, Mehta S, Verma A, Gothwal S, Goudar SS, Derman R, Katheria A, Aghai ZH. CORDMILK: Umbilical Cord Milking versus Early Cord Clamping on short-and long-term outcomes in neonates who are non-vigorous at birth-study protocol of a multi-center, cluster-randomized, crossover-controlled trial. Trials. 2025 Nov 17;26(1):509. doi: 10.1186/s13063-025-09197-8. PMID 41250198